CLINICAL TRIAL: NCT00908570
Title: Topical Estriol for Vaginal Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: University of Illinois at Chicago (Other); University of California, Los Angeles (Other); Tulane University School of Medicine (Other); Magee-Women's Research Institute (Other); Oregon Health and Science University (Other)
Responsible Party: Beverly Winikoff, MD, MPH, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5.1
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Vaginal Health
Keywords: estrogen; estriol; cream; vagina; infection prevention
MeSH Terms: interventions — Estriol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1Topical estriol cream (Experimental)
  Interventions: Drug: estriol
- 2Placebo cream (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: estriol — 4 ml vaginal cream (1.0 mg estriol/1 ml cream), 3 days/week for approximately 2 months.
  Arms: 1Topical estriol cream
Drug: Placebo — Placebo cream
  Arms: 2Placebo cream

SUMMARY:
The purpose of this Phase I study is to investigate and document the effects of local treatment with a topical estriol cream on the vaginal environment of pre-menopausal women.

DETAILED DESCRIPTION:
There is evidence from human studies that estrogen can give rise to health-promoting changes in the vaginal environment in addition to affecting the thickness of the vaginal epithelium. The purpose of the proposed study is to take the first steps in testing the effects of local estrogen treatment on vaginal health parameters in humans. We have chosen an estriol product because, in comparison with estrone (E1) and estradiol (E2), estriol (E3) is generally considered to be a weak estrogen. The duration of estriol's interaction with the estrogen receptor is quick and exhibits rapid metabolic clearance. We have chosen a topical route of administration because it appears to result in fewer systemic effects than oral administration, while allowing us to concentrate treatment locally in the areas we wish to affect.

Our primary goal is to test whether or not topically applied estrogen results in significant thickening and maturation of the vaginal epithelium. Our secondary goal is to measure the treatment's effects on other parameters of the vagina, such as Lactobacillus colonization and vaginal pH. If estrogen cream does indeed affect the vaginal environment in pre-menopausal women as it does in post-menopausal women, further study would be indicated to determine whether estrogen cream in the vagina decreases risk of infection in pre-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* In generally good health
* Between the ages of 18 and 40
* Report regular, consistent menstrual cycles with duration between 25 and 35 days' duration
* Agree not to initiate hormonal contraception or other systemic or vaginal hormonal treatments during the course of the study
* Agree to refrain from vaginal douching and use of spermicides, spermicide-treated condoms, diaphragms, cervical caps, vaginal hygiene treatments and other vaginal products during the course of the study except as explicitly allowed under study protocol.
* Not attempting to get pregnant (and, if sexually active, using an allowed effective contraceptive - i.e., sterilization or male condoms)

Exclusion Criteria:

* Has been informed by a health practitioner that she should avoid estrogen treatments
* Does not meet one or more of the above inclusion criteria
* Is currently pregnant
* Is currently lactating
* Has IUD in place
* Has diabetes that is controlled with medication
* Has menstrual bleeding that usually exceeds 7 days' duration
* Has used hormonal contraception or other systemic or vaginal hormonal treatment during the past three months
* Has received systemic antibiotic treatment since the start of bleeding in her current menstrual period
* Has known history of diagnosis of HIV infection
* Screens positive for gonorrhea, Chlamydia, or trichomonas
* Has evidence of high-grade dysplasia or cervical cancer on visual examination or Pap smear
* Has active genital Herpes lesions
* Has any of the following:
* Known, past or suspected breast cancer;
* Known or suspected estrogen-dependent malignant or pre-malignant tumours (e.g endometrial cancer);
* History of endometrial hyperplasia;
* Undiagnosed or abnormal genital bleeding;
* Previous idiopathic or current venous thromboembolism (deep venous thrombosis, pulmonary embolism);
* Active or recent arterial thromboembolic disease (e.g. angina, myocardial infarction);
* Acute liver disease, or a history of liver disease where liver function tests have failed to return to normal;
* Liver disorders such as adenomas;
* Symptomatic gallstones or gallbladder disease (cholecystitis);
* Hypertriglyceridemia;
* Vascular disease associated with lupus erythematosus;
* Known hypersensitivity to estriol (estrogen E3) or the inactive substances in the study product;
* Porphyria
* Presents any other history or condition that provider, in his or her best discretion, feels should rule out study participation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in thickness of the vaginal epithelium | Pre and post treatment luteal and follicular phases

SECONDARY OUTCOMES:
Other vaginal parameters including Lactobacillus colonization and vaginal pH | Pre and post treatment follicular and luteal phases

CONTACTS AND LOCATIONS:
Overall Officials: Yael Swica, M.D., M.P.H., Principal Investigator — Gynuity Health Projects
Locations (2):
- United States (2):
  - Harbor-UCLA Medical Center, Los Angeles, California
  - University of Illinois at Chicago, Chicago, Illinois